CLINICAL TRIAL: NCT01039038
Title: A Phase II Study Evaluating the Feasibility of a Dose Increase by a Boost of Curietherapy in PDR Associated With the Extern Radiotherapy in Intermediate Risk in the Prostate Cancer
Brief Title: Feasibility Study of a Dose Increase by a Boost of Curietherapy in Pulse Dose Rate (PDR) Associated With the Extern Radiotherapy in Prostate Cancer
Acronym: CURIEBOOST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Dr Anne-Catherine COURTECUISSE-DEGRENDEL, Centre François Baclesse
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CURIEBOOST
Record Dates: First submitted 2009-12-11; First posted 2009-12-24 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Prostate Cancer With Intermediate Risk
Keywords: prostate; curietherapy; radiotherapy; intermediate risk
MeSH Terms: interventions — Brachytherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: curietherapy and radiotherapy — boost of curietherapy(40 Gy)and external radiotherapy (34 Gy)

SUMMARY:
The objective of the trial is to evaluating the feasibility of dose increase by a boost of curietherapy in PDR (at least 40 Gy on D95) associated to extern radiotherapy (34 Gy) in intermediate risk in prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years and ≤ 75 years
* Life expectancy >10 years
* Localized prostatic adenocarcinoma and histologically proven
* Intermediate risk cancer(T2b or PSA between 10 and 20 or Gleason = 7(3+4) according to Amico criteria
* Metastasis or pelvic pathologic ganglion (≥ 10 mm) absence
* OMS < 2
* No previous treatment by radiotherapy and/or curietherapy
* Hormonotherapy authorized before and during the study
* Rectal or uretero-vesical pathology
* Signed informed consent
* Social security system affiliation
* Individual deprived of liberty or placed under the authority of a tutor.
* No anesthesia contraindication

Exclusion Criteria:

* Adenocarcinoma not histologically proven
* Metastases presence
* Pathological nodes presence(≥ 10 mm)
* Prior prostate endoscopic resection
* history of other malignancy except for appropriately treated superficial basal cell skin cancer
* Medical contraindications to anesthesia
* Patients with uncontrolled psychiatric disease or medical disease incompatible with the protocol
* Impossibility to respect the medical follow-up of the protocol for geographical, social or psychic reasons

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a delivered dose by a boost of curietherapy is at least 40 Gy (D95) associated to a dose of 34 Gy for extern radiotherapy | at 5 months

SECONDARY OUTCOMES:
Acute toxicities at month 3 after end of treatment: late toxicities, survival without biological relapse, without local relapse or metastatic evolution, feasibility of MRI use in prostatic CTV | at 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, Basse-normandie, France